CLINICAL TRIAL: NCT03409432
Title: A Phase II Study of Brentuximab Vedotin and Lenalidomide in Relapsed and Refractory T-Cell Lymphomas
Brief Title: Brentuximab Vedotin and Lenalidomide in Treating Patients With Stage IB-IVB Relapsed or Refractory T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Reneau (Other)
Responsible Party: Sponsor-Investigator, John Reneau, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17204; NCI-2017-02221 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-04; First posted 2018-01-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Lymphomatoid Papulosis; Primary Cutaneous Anaplastic Large Cell Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage I Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage II Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage III Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage IV Cutaneous T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphomatoid Papulosis; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell | interventions — Brentuximab Vedotin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brentuximab vedotin, lenalidomide) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 and lenalidomide PO QD on day 1-21. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies how well brentuximab vedotin and lenalidomide work in treating patients with stage IB-IVB T-cell lymphoma that have come back or do not respond to treatment. Monoclonal antibodies, such as brentuximab vedotin, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving brentuximab vedotin and lenalidomide may work better in treating patients with T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) of the combination of brentuximab vedotin (BV) and lenalidomide in patients with relapsed or refractory cutaneous T-cell lymphoma (CTCL)/peripheral T-cell lymphoma (PTCL).

SECONDARY OBJECTIVES:

I. To estimate the duration of response and 2 year progression-free survival (PFS) and overall survival (OS) associated with the combination of brentuximab vedotin (BV) and lenalidomide in patients with relapsed or refractory CTCL/PTCL.

II. To define the qualitative and quantitative toxicities of the combination of brentuximab vedotin (BV) and lenalidomide in patients with relapsed or refractory CTCL/PTCL.

TERTIARY OBJECTIVES:

I. To correlate between the expression of CD30 in neoplastic cells by immunohistochemistry (IHC) and overall response rate (ORR) of the combination of brentuximab vedotin (BV) and lenalidomide in patients with relapsed or refractory CTCL/PTCL.

II. To determine T-cell and natural killer (NK) cell subset numbers, phenotype, and functional status in relapsed or refractory (rel/ref) CTCL/PTCL patients, and whether the combination of brentuximab vedotin and lenalidomide alters these parameters during therapy.

III. To determine changes in plasma cytokine levels and other biomarkers in this patient population during therapy with the combination of brentuximab vedotin and lenalidomide.

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1 and lenalidomide orally (PO) once daily (QD) on day 1-21. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Biopsy-proven, measurable, stage IB-IVB relapsed or refractory cutaneous T-cell lymphoma after 2 lines of skin-directed therapy or one prior line of systemic therapy

  * (Note: extracorporeal photopheresis will be considered a systemic therapy for this study)
* Patients with large cell transformation of cutaneous T cell lymphoma are eligible
* Patients with advanced stage non-mycosis fungoides (MF) CTCL are eligible including, but not limited to, advanced stage lymphomatoid papulosis (LyP) or primary cutaneous anaplastic large cell lymphoma (pcALCL)
* Patients with systemic T cell lymphoma of any stage and any subtypes; patient must have had at least one standard chemotherapy and measurable disease at the time of enrollment; bidimensional measurable disease of at least 1.5 cm in the greatest transverse diameter as documented by computed tomography (CT) or positron emission tomography (PET)/CT
* Patients with systemic T cell lymphomas who relapsed after autologous transplant are eligible
* Prior treatment with brentuximab vedotin is allowed provided the patient did not progress on BV or within 30 days of last dose of BV; patients must be at least 3 months from the last dose of BV
* CD30 staining is to be performed on fresh biopsy or archival formalin-fixed paraffin-embedded (FFPE) tissue however CD30 positivity is not required for eligibility
* All cancer therapy, including radiation, topical steroid, and chemotherapy must have been discontinued at least 1 week or 3 half-lives whichever is the longest prior to treatment in this study; the only exceptions are participants who are symptomatic from their skin lesions and have been on corticosteroids for prolonged periods of time (> 60 days) without change may continue use of either systemic steroids (equivalent to < 10 mg per day of prednisone) or topical steroids are eligible for this study if the frequency and dosage steroids has not changed for 60 days prior to the study; these participants should continue on the same dose of systemic/topical steroid throughout the study period unless they achieve a complete response at which time steroids can be discontinued; patients are allowed to continue any medications with known activity in T cell lymphomas at the pre-enrollment doses for conditions other than T cell lymphomas (ie, steroids for sarcoidosis), as long as there is evidence of T cell lymphoma progression while patients were on these agents
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Absolute neutrophil count >= 1000/mm^3
* Platelet count >= 50,000/mm^3
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* AST (SGOT) and ALT (SGPT) =< 5 x ULN in patients with documented hepatic involvement by lymphoma
* Calculated creatinine clearance >= 60 ml/min (by the Cockcroft-Gault equation)
* Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast; patients with early stage of prostate cancer under clinical surveillance without therapy are eligible
* Negative serum pregnancy test at the time of enrollment for females of childbearing potential
* Women of childbearing potential must follow pregnancy testing requirements as outlined in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program material; this is defined as either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of contraception (one highly effective method and one additional effective method (AT THE SAME TIME) at least 28 days prior to the start of lenalidomide, for the duration of study participation, and for 28 days following the last doses of brentuximab vedotin and lenalidomide; women of childbearing potential must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a woman of childbearing potential even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* All study participants must be registered into the mandatory Revlimid REMS program and be willing to comply with its requirements; per standard Revlimid REMS program requirements, all physicians who prescribe lenalidomide for research subjects enrolled into this trial, must be registered in, and must comply with, all requirements of the Revlimid REMS program
* Life expectancy > 30 days

Exclusion Criteria:

* Patients with active central nervous system (CNS) involvement with lymphoma are not eligible
* Patients with pre-existing grade >= 3 peripheral neuropathy
* Patients with known human immunodeficiency virus (HIV) infection or are not eligible
* Patients who had solid organ transplants are not eligible
* Evidence of active hepatitis B infection, based on positive surface antigen or hepatitis B deoxyribonucleic acid (DNA) polymerase chain reaction (PCR), or active hepatitis C infection; patients who are hepatitis B core antibody positive must take prophylaxis with lamivudine or equivalent and be willing to undergo monthly hepatitis B DNA PCR testing
* Present or history of progressive multifocal leukoencephalopathy (PML)
* Prior allogeneic stem cell transplant is not permitted
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction likely to interfere with the delivery, absorption, or metabolism of lenalidomide
* Patients may take steroids for disease control up to 24 hours prior to study enrollment; topical steroids are allowed for CTCL patients as described in inclusion criteria above
* Any illness, medical condition or organ system dysfunction which, in the investigator?s opinion, could compromise the subject?s safety, interfere with the absorption or metabolism of lenalidomide, or put the study outcomes at undue risk
* A cardiovascular disability status of New York Heart Association class >= 2
* History of severe allergic reactions to humanized monoclonal antibodies
* History of other malignancy that could affect compliance with the protocol or interpretation of results; patients with a history of curatively treated basal or squamous cell carcinoma or stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible; individuals in documented remission without treatment for 2 years prior to enrollment may be included at the discretion of the investigator; patients with early stage of prostate cancer under clinical surveillance without therapy are eligible
* Known hypersensitivity to any of the study drugs or analogs
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior study therapy
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Recent major surgery (within 6 weeks prior to the start of study treatment) other than for diagnosis
* Receiving immunosuppressive therapy
* Refractory to prior therapy with brentuximab vedotin (evidence of progression within 30 days of the last dose)
* Prior therapy with lenalidomide
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years
  the overall response rate (ORR) of the combination of brentuximab vedotin (BV) and lenalidomide in patients with relapsed or refractory CTCL/PTCL

SECONDARY OUTCOMES:
Incidence of adverse events according to National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days after last day of study treatment
  Toxicity will be graded by the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0
Overall survival (OS) | From start of study treatment to date of death due to any cause, assessed up to 2 years
  Kaplan-Meier method will be used to estimate OS.
Progression free survival (PFS) | From start of study treatment to first documentation of tumor progression (including radiographic and clinical progression) or to death due to any cause, whichever comes first, assessed up to 2 years
  Kaplan-Meier method will be used to estimate PFS.

CONTACTS AND LOCATIONS:
Overall Officials: John Reneau, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu